CLINICAL TRIAL: NCT01802658
Title: Bone Demineralization Lesions in the Injured Marrow: Efficacy and Tolerability of Administration Early and Repeated the Zoledronic Acid. Comparative Study, Prospective, Double-blind Controlled
Brief Title: Bone Demineralization Lesions in the Injured Marrow: Efficacy and Tolerability of Administration Early and Repeated the Zoledronic Acid. Comparative Study, Prospective, Double-blind Controlled (DBMZol)
Acronym: DBMZol
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruiting Difficulty
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRD/11/06-P; 2012-001778-27 (EudraCT Number)
Record Dates: First submitted 2013-02-28; First posted 2013-03-01 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Bone Demineralization Lesions in the Injured Marrow
Keywords: Bone marrow demineralization lesions,: efficacy and tolerability, zoledronic acid
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic acid (Active Comparator): Zoledronic acid 5 mg. IV. 3 infusions. Administration 3 times over two years.
  Interventions: Drug: Zoledronic acid
- NACL (Placebo Comparator): NACl 100 ml IV. 3 infusions. Administration 3 times over two years.
  Interventions: Drug: NA Cl

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid 5 mg. IV. 3 infusions. Administration 3 times inclusion M12 and M24 over two years.
  Arms: Zoledronic acid
Drug: NA Cl — NACl 100 ml IV. 3 infusions. Administration 3 times inclusion M12, M24 over two years.
  Arms: NACL

SUMMARY:
Subjects with lesion bone marrow are at risk of fracture by fragility bone. The median time to onset of fracture was 8.5 years. Fracture increases costs of care, dependency.

Bone fragility is secondary to hormonal disorders and calcium phosphate, impaired excretion of neuropeptides, vasomotor symptoms associated with the asset that promote bone loss and architectural disorganization. These phenomena occur in the first weeks of development of spinal cord injury and predominate in the distal femur and proximal tibia. From the third year, the demineralization stabilizes, bone mass is estimated to be between 70 and 50% of the initial bone mass, the new equilibrium.

No clinical evidence is predictive of fracture risk. A criteria surrogate must be used to assess this risk. There is an association between bone mineral density and fracture risk. The fracture threshold knee was evaluated to 0.87 g/cm2. Evaluation of bone mineral density in the distal femur is a predictor of fracture risk. Measure reliable and reproducible, easy to perform, it is a good element for monitoring the efficacy of anti-resorptive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with a spinal cord injury less than 12 weeks of etiology stable,
* level of injury C5 L2,
* AIS grade A to D.
* Female or male between 18 and 45 years.
* No pregnancy.
* No osteoporosis.
* Good oral health.
* Good glomerular filtration.
* No cons-indication to Zoledronic Acid.
* No drugs affecting bone metabolism

Exclusion Criteria:

* pregnancy.
* osteoporosis.
* cons-indication to Zoledronic Acid.
* drugs affecting bone metabolism

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
determine DMO distal femur at 36 months | october 2015

SECONDARY OUTCOMES:
Incidence of fractures of members lower in the first 36 months. | october 2015
  to determine incidence of fractures of members lower in the first 36 months
Response to the EQ-5D questionnaire at baseline, M12, M24, M36. | october 2015
  To determine the EQ-5D
DMO (g/cm2) at the distal femur, proximal femur, spine, total body M6, M12, M24, M36. | october 2015
  Determine the DMO
Bioassays: b CTX, PAO, PINP at M6, M12, M24, M36 | october 2015
  to measure bioassays

OTHER OUTCOMES:
Further study of biological markers of bone resorption | october 2015
Study of bone architecture by QCT p | october 2015
Establishment of a bio-collection. | october 2015
Additional clinical follow-up study. | october 2015
Medico-economic analysis. | october 2015

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Centre Bouffard - Vercelli CAP Cerbère, Cervera de la Marenda
  - CRMPR Les Herbiers, Les Herbiers
  - Centre Mutualiste Neurologique Propara, Montpellier
  - Institut Régional de Réadaptation Nancy, Nancy
  - University hospital of Nantes, Nantes
  - Hôpital R. Poincaré, Paris
  - CHU, Saint-Etienne
  - Centre de l'Arche, Saint-Saturnin
  - Hôpital Rangueil CHU, Toulouse